CLINICAL TRIAL: NCT00675077
Title: Phase 1 Study to Determine the Efficacy of Using Far Infrared Radiation for Control, Management and Treatment of HD
Brief Title: Far Infrared Irradiation for Managing, Control and Treatment of Huntington's Disease (HD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-HD-CTP1
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Huntington Disease
Keywords: Akinetic-Rigid Variant of Huntington Disease; Chorea, Chronic Progressive Hereditary (Huntington); Chronic Progressive Hereditary Chorea (Huntington); Huntington Chorea; Huntington Chronic Progressive Hereditary Chorea; Huntington Disease, Akinetic-Rigid Variant; Huntington Disease, Juvenile; Huntington Disease, Juvenile-Onset
MeSH Terms: conditions — Huntington Disease; Chorea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Radiation: Far Infrared Radiation (5μm to 20μm wavelength)
  Interventions: Radiation: Far Infrared Radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation — Far Infrared Radiation (5μm to 20μm wavelength). Far Infrared radiation for 30 to 40 minutes per treatment session.
  Other Names: Far Infrared Radiation (5μm to 20μm wavelength)

SUMMARY:
Huntington's disease (HD) is a fatal disease with profound neurological and behavioral features. HD is typically characterized by uncontrollable movements and psychological disturbances.

This study will investigate the use of far infrared radiation for control, management and treatment of HD.

DETAILED DESCRIPTION:
Observations from our research studies indicate that, far infrared rays provide energy to the body, improve the autonomic functions of the nervous system, restore the functions of the endocrine system, strengthen the immune system, improve blood circulation and increase the level of oxygen in the cells and promote the regeneration of muscle cells, nerves and brain cells.

It is hereby postulated that irradiation using far infrared, with wavelength between 5 to 20 microns, of the central nervous system, the endocrine system and the whole body could prevent, control, manage or possibly lead to complete rehabilitation of people who have HD.

ELIGIBILITY:
Inclusion Criteria:

* People with HD

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Treatment of people with HD | 2 years

SECONDARY OUTCOMES:
Rehabilitation of people with HD | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada